CLINICAL TRIAL: NCT05620446
Title: Endoscopic Management of Acute Sigmoid Volvulus in High Risk Surgical Eldery Patients: A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ahmed Shafiq
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Elderly Patient Withsigmoid Volvulus
Keywords: endoscopic surgery
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled clinical trial included all patients who developed the manifestations of acute a cute sigmoid volvulus and referred to the Zagazig University Hospital Emergency Department between December 2020 and August 2022. The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 9989/23-10-2022), Included eligible patients were simply randomized at a 1:1 ratio to "Endoscopic (SG)" or "Surgical Colostomy Group (EG)" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic managment of sigmoid volvulus (Active Comparator): patients are subjected to untwist the volvulus first by endoscopy then one or two days later are subjected to sigmoid colon fixation by endoscopy using 2-shot anchor device
  Interventions: Procedure: endoscopy
- surgical management of sigmoid volvulus (No Intervention): patients aresubjected for surgical colostomy ( hartman's procedure ) , then later on after 6 weeks , they are subjected for surgical sigmoid fixation or excision either by open or laparoscopic approach

INTERVENTIONS:
Procedure: endoscopy — the technique was done by two doctor the patients were sedated then colonoscopy was done for the patients while the patients were put in lithotomy position , we identified the site of sigmoid colon fixation by radiological colongraphy then tip of artery forceps was moved at outer skin at anterior abdominal wall at left lower quadrant to meet tip of colonscopy at multiple point where fixation was done . fixation was done by exploratory puncture of skin by scalpel about (2-3 mm puncture) at site of these points then widening the puncture by artery forceps at level of subcutaneous tissue. A 2- shot anchor device was used to fix the sigmoid colon against anterior abdominal wall. The 2-shot anchor device was passed through the puncture to be entered inside the sigmoid colon and the thread with a metal T-bar was detachd and pulled towards the anterior abdominal wall. This was repeated at multiple point of fixation .
  Arms: endoscopic managment of sigmoid volvulus

SUMMARY:
This prospective randomized controlled clinical trial included all patients who developed the manifestations of acute a cute sigmoid volvulus and referred to the Zagazig University Hospital Emergency Department between December 2020 and August 2022. The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 9989/23-10-2022), Patients with age of ≥60 years-old , with acute sigmoid volvulus not managed by rectal deflating tube, with no evidence of bowel ischemia, with ASA III & IV , high risk surgical patients , with comorbidities and on sepsis but not septic shock were included and eligible for randomization. We excluded patients who were with good general condition (ASAI&II), patients with age below 60 years , patients with bowel ischemia and patients managed by rectal deflating tube.

Included eligible patients were simply randomized at a 1:1 ratio to "Endoscopic (SG)" or "Surgical Colostomy Group (EG)" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.

DETAILED DESCRIPTION:
Introduction:

Sigmoid volvulus is a surgical emergency and if untreated, it will lead to bowel ischemia & perforation with high incidence of mortality (1). Most of the patients with sigmoid volvulus are old age with many co-morbidities (2). So, the risk of surgery for those elderly patients is high and is associated with high incidence of morbidity & mortality (3) . Early intervention is required for managing the sigmoid volvulus to avoid its serious complications , so the less invasive intervention is the best for those high risk elderly patients (4) . Usually in the past after failure of deflating rectal tube to untwist the volvulus , the patients were subjected for surgical colostomy to relive the intestinal obstruction with high risk consent for elderly patients then in later session , they were subjected for definitive surgery (5) . As the emergency surgery is associated with high incidence of morbidity & mortality in elderly patients, so the endoscopic approach becomes the first line of management to resolve the obstruction in uncomplicated sigmoid volvulus in elderly patients (6). The endoscopic untwist of the acute sigmoid volvulus was first described by Bruusgaard and had the advantage of both diagnostic & therapeutic values (7) . For diagnostic value, the endoscopy evaluate the mucosa and its viability , it is also important to exclude other causes of intestinal obstruction , the length of the endoscopy is enough to reach beyond site of twist and diagnose the torsion as the site of twist appears spiral , sphincter area of the mucosa (8). For therapeutic value , it is successful in treating the acute volvulus by incidence of 75%-95% , but with high recurrence rate up to 90% (9). The elective definitive surgery few days later after the endoscopy was postponed in elderly patients for many reasons , so in our study we will try to fix the sigmoid colon also by endoscopy without needs for general anesthesia and major surgery.

Objectives:

To evaluate the advantages and safety of Endoscopic management of acute sigmoid volvulus in high risk surgical patients and its effect in reducing morbidity and postoperative hospital stay.

Patients and Methods Patients This prospective randomized controlled clinical trial included all patients who developed the manifestations of acute a cute sigmoid volvulus and referred to the Zagazig University Hospital Emergency Department between December 2020 and August 2022. The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 9989/23-10-2022), and was retrospectively submitted in clinicaltrials.gov in November 2022 (NCT05051683). The study was performed in accordance with the code of ethics of the World Medical Association (Declaration of Helsinki) for studies involving human subjects. Written informed consent was obtained from all participants after explaining to them all the study procedures with its benefits and hazards. Patients with age of ≥60 years-old , with acute sigmoid volvulus not managed by rectal deflating tube, with no evidence of bowel ischemia, with ASA III & IV , high risk surgical patients , with comorbidities and on sepsis but not septic shock were included and eligible for randomization. We excluded patients who were with good general condition (ASAI&II), patients with age below 60 years , patients with bowel ischemia and patients managed by rectal deflating tube.

Included eligible patients were simply randomized at a 1:1 ratio to "Endoscopic (SG)" or "Surgical Colostomy Group (EG)" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.

The sample size was calculated by using open Epi program depending on the following data ; confidence interval 95% , power of the test 80% , ratio of unexposed/ exposed 1 , the success rate of surgical colostomy versus endoscopic colostomy was 90 % versus 15% respectively. Odd ratio 0.02 , and risk ratio 0.17 , so the calculated sample size equal 18 patients divided into two equal groups. Primary and secondary outcomes were success rate in managing the obstruction , postoperative hospital stay, and complications and mortality in each group after the intervention during the 3-months follow-up period, respectively.

Diagnosis After full history taking and complete physical examination, acute sigmoid volvulus was clinically suspected and then confirmed by laboratory investigations (complete blood picture, liver and kidney functions, coagulation profile), radiological imaging (plain erect chest X-ray abdomen, abdominal US , CT abdomen with oral and I.V contrast and virtual colonscopy ).

Intervention:

For group A ( endoscopy group ): after admission of the patients to the emergency department & confirmation of the diagnosis , the included patients in this group were subjected for rapid resuscitation in ICU or inpatient bed according to patient's general condition then rapidly were subjected for colonoscopy under sedation in operative room to untwist the volvulus by passing the colonoscopy (CF260 series; Olympus, Tokyo, Japan) to site of volvulus which was appeared as spiral & sphincter area of the mucosa . The untwist was done under radiological guidance of C-arm by gas suction & insufflation till untwisting was occurred . Then rectal tube was put to avoid recurrence of volvulus and also for washing & irrigation of the colon by ringer or saline solution ( 500cc /8h for one or two days ) at inpatient bed or ICU bed according to patient's general condition to get the colon empty from stool. After that patients ( after one or two days ) the patients were shifted again to operative room for sigmoid colon fixation by endoscopy as following : the technique was done by two doctor ( one for endoscopy and the other for sigmoid fixation ) the patients were sedated after intravenous preoperative ceftriaxone & metronidazole injection , then colonoscopy was done for the patients while the patients were put in lithotomy position , we identified the site of sigmoid colon fixation by radiological colongraphy by injection of radio-opaque dye via the endoscopy then tip of artery forceps was moved at outer skin at anterior abdominal wall at left lower quadrant to meet tip of colonscopy at multiple point where fixation was done ( at least 4 to 5 points of fixation ) . fixation was done by exploratory puncture of skin by scalpel about (2-3 mm puncture) at site of these points then widening the puncture by artery forceps at level of subcutaneous tissue. A 2- shot anchor device ( Olympus, Tokyo , Japan) was used to fix the sigmoid colon against anterior abdominal wall. After exploratory puncture was done , a 20-gauge needle was used for further confirmation of site of fixation. A suction test was performed to exclude presence of intervening organ between sigmoid colon and anterior abdominal wall. The 2-shot anchor device was passed through the puncture to be entered inside the sigmoid colon and the thread with a metal T-bar was detached and pulled towards the anterior abdominal wall. This was repeated at multiple point of fixation (4-5 points of fixation ). Ct-colongraphy ( virtual colongraphy ) was done on next day at morning before patient's discharge to confirm sigmoid fixation and avoid missing any leak .

For group B ( surgical group ) : after admission of the patients to the emergency department & confirmation of the diagnosis , the included patients in this group were subjected for rapid resuscitation in ICU or inpatient bed according to patient's general condition then rapidly were subjected for surgical colostomy ( hartman's procedure ) , then later on after 6 weeks , they were subjected for surgical sigmoid fixation or excision either by open or laparoscopic approach . In this group , the patients were discharged after colostomy then readmission again after 6 weeks for definitive surgery.

Statistical analysis Analysis of data was performed using SPSS (Statistical Package of Social Services) version 22. Quantitative variables were described as mean (±SD, standard deviation) and median (range) according to Shapiro test of normality. Qualitative variables were described as a number and a percent. Chi-square test was used to compare qualitative variables between the 2 groups. Fisher exact test was used when one expected cell or more are less than 5. Unpaired t-test was used to compare quantitative variables, in parametric data (SD < 30% of the mean). Mann Whitney test was used instead of unpaired t-test in non-parametric data (SD > 30% of the mean). The results were considered statistically significant when the significant probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically significant (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS)(10).

ELIGIBILITY:
Inclusion Criteria:

* Patients with age of ≥60 years-old ,
* patients with acute sigmoid volvulus not managed by rectal deflating tube,
* patients with no evidence of bowel ischemia,
* patients with ASA III & IV , high risk surgical patients ,
* patientswith comorbidities
* patients on sepsis but not septic shock

Exclusion Criteria:

* patients with good general condition (ASAI&II),
* patients with age below 60 years ,
* patients with bowel ischemia
* patients managed by rectal deflating tube

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
efficacy and safety of endoscopic management of acute sigmoid volvulus | within one week after intervention
  incidence of postoperative complication

SECONDARY OUTCOMES:
efficacy of endoscopic management of acute sigmoid volvulus | within 6 month post operative
  incidence of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — Zagazig University Hospitals
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Negm S, Farag A, Shafiq A, Moursi A, Abdelghani AA. Endoscopic management of acute sigmoid volvulus in high risk surgical elderly patients: a randomized controlled trial. Langenbecks Arch Surg. 2023 Aug 28;408(1):338. doi: 10.1007/s00423-023-03071-4. PMID 37635200